CLINICAL TRIAL: NCT05040685
Title: Axillary Reverse Mapping (ARM): Validation of Surgical Tecnique in Breast Cancer Surgery
Brief Title: Axillary Reverse Mapping in Breast Cancer
Acronym: ARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR139/21
Record Dates: First submitted 2021-08-19; First posted 2021-09-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Lymph Node Cancer Metastatic
Keywords: Lymphedema; Sentinel lymph node; Axillary lymph node dissection
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: This is a prospective not randomized pilot study to validate the axillary mapping reverse technique by using indocyanine green.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axillary mapping reverse (Experimental): Application of axillary mapping reverse technique
  Interventions: Procedure: Axillary mapping reverse

INTERVENTIONS:
Procedure: Axillary mapping reverse — At the time of performing the ALND associate the ARM, injecting between 2-5mL of indocyanine green subcutaneously in the ipsilateral upper extremity at the medial inter-muscular and massaged for 5 min. First, identify the ARM nodes by indocyanine green, then perform conventional axillary lymphadenectomy trying to preserve the ARM nodes. And, in a second time, extract ARM nodes for their individualized anatomopathological study.

SUMMARY:
The axillary mapping reverse (ARM) consists in differentiating the upper limb lymph nodes from the breast ones in order to preserve them and reduce the possibility of lymphedema.

A significant decrease of lymphedema rates in patients who was possible associate ARM technique during the axillary surgery improving the quality of life of these patients. There are different visualisation techniques like fluorescence dye.

DETAILED DESCRIPTION:
Axillary lymph node dissection (ALND) was the standard therapy until 1990-2000, when the technique was replaced, when possible, by another procedure associated with less morbidity: the sentinel lymph node biopsy (SLNB). However, actually, ALND is still the gold standard in some patients. This procedure is associated with substantial morbidity, like lymphedema, shoulder pain, arm numbness, axillary web syndrome and decreased upper-extremity range of motion (ROM), that severely conditions the quality of life of these patients.

In 2007, the investigators had the first reports about a new surgical technique, the axillary mapping reverse (ARM), that consists in differentiating the upper limb lymph nodes from the breast ones in order to preserve them and reduce the possibility of lymphedema.

The current literature shows a significant decrease of lymphedema rates in patients who was possible associate this technique during the axillary surgery improving the quality of life of these patients. There are different visualisation techniques. With the use of indocyanine green, the visualisation rates in the axilla of ARM lymphatics are from 88%, similar to other techniques. Some advantages of fluorescence dye are that no systemic allergic reactions have been reported and the 'green tattoo' disappears quickly.

HYPHOTESIS The axillary mapping reverse (AMR) is able to identify the lymph nodes responsible for lymphatic drainage of the ipsilateral upper limb (ARM nodes) in breast cancer patients who underwent an axillar lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

Patients who will undergo ALND in the treatment of breast cancer:

* cT4a, cT4c and cT4d.
* cT4b with extensive involvement of the skin.
* cN0 with SLNB positive (pN+) that need to associate ALND:

  * cT3-T4b.
  * >2 lymph node macrometastasis if cTis, cT1 and cT2.
  * Patients who underwent mastectomy and it is not possible associate adjuvant radiotherapy.
* cN1:

  * If primary surgery treatment.
  * After neoadjuvant systemic treatment, if there is not a clinical-radiological complete response and/or SLNB positive (ypN+).
* cN2:

  * If primary surgery treatment.
  * After neoadjuvant systemic treatment, if luminal tumours or there is not a clinical-radiological complete response in triple negative or HER2 overexpressed tumours.
* cN3.

Exclusion Criteria:

* Patients with previous axillary surgery (except sentinel node biopsy)
* Patients who did previous axillary radiotherapy treatment.
* Patients who do not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of patients who it is possible preserve ARM nodes | 1 year
  Determinate the percentage of patients who is possible preserve the ARM node during ALND

SECONDARY OUTCOMES:
Rate of metastatic ARM | 1 year
  Determinate the percentage of metastatic ARM nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ortega Expósito, MD, Principal Investigator — Bellvitge Hospital
Locations (1):
- Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No